CLINICAL TRIAL: NCT06544148
Title: Non-Invasive Measurements of Changes in Pulmonary Artery Pressure in Intensive Care Unit Patients Using Electrical Impedance Tomography - A Feasibility Study (PAP-EIT Study)
Brief Title: Non-Invasive Measurements of Changes in Pulmonary Artery Pressure in Intensive Care Unit Patients Using Electrical Impedance Tomography - A Feasibility Study
Acronym: PAP-EIT
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-00435
Record Dates: First submitted 2024-07-22; First posted 2024-08-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Study Participants
  Interventions: Device: Electrical impedance tomography

INTERVENTIONS:
Device: Electrical impedance tomography — In addition to routine critical care with a pulmonary artery catheter already in place (PAC), an electrical impedance tomography (EIT) belt will be placed in patients enrolled in this study. Data will be analyzed offline and clinical trajectory and/or decisions will not be impacted by this additional monitoring. EIT is a non-invasive, safe, and radiation-free medical imaging modality.

SUMMARY:
To assess whether changes in electrical impedance - measured using an electrical impedance tomography (EIT) chest belt - can be used to derive changes in pulmonary artery pressure (PAP) in critically ill patients when compared to invasive gold-standard PAP measured using pulmonary artery catheter (PAC).

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18-year-old.
* Intubated patients in the ICU with clinical decision to monitor PAP and cardiac output using a PAC.

Exclusion criteria:

* Patients with implanted or external thoracic electronic devices (e.g., pacemaker) or thoracic metal implants.
* Known pregnancy or lactating patients.
* Open lung injuries or pneumothorax.
* Open wounds, drainages, burns or rashes of the upper thorax.
* Estimated thoracic perimeter smaller than 66 cm or larger than 134 cm.
* Known allergies to wound dressings or adhesives (e.g., gel electrodes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study the investigators plan to enroll 28 patients with complete datasets for evaluation of PAP derived by PAC and EIT for a minimum duration of 4 hours in the ICU at Inselspital (Bern) with clinical decision to monitor PAP using a PAC.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2027-08-05 (Estimated)

PRIMARY OUTCOMES:
Mean difference between EIT-derived and PAC-measured changes in pulmonary artery pressure | Up to 48 hours
  The primary outcome is the difference - expressed as mean and standard deviation (SD) - between changes in EIT-derived pulmonary artery pressure (ΔPAP_EIT), derived from changes in the pulmonary pulse arrival time, and changes in pulmonary artery catheter-based pulmonary artery pressure (ΔPAP_PAC). This will be measured over recording periods of up to 48 hours.

SECONDARY OUTCOMES:
Data acceptance rate | Up to 48 hours
  Data acceptance rate, i.e., the percentage of total recording duration during which lung EIT signals show pulmonary pressure morphology and thus allow to estimate EIT-derived PAP values.
Concordance rate (%) of directional changes in pulmonary artery pressure between EIT and PAC measurements (Trending ability) | Up to 48 hours
  The trending ability will be assessed using four quadrant plot analysis to calculate the concordance rate between EIT-derived and PAC-measured pulmonary artery pressure changes. The concordance rate is defined as the percentage of data points in which both methods agree on the direction of change (increase or decrease) in pulmonary artery pressure.
Accuracy and trending ability of EIT-derived cardiac output compared to PAC measurements | Up to 48 hours
  The difference between EIT-derived cardiac output (CO_EIT) and pulmonary artery catheter-based cardiac output (CO_PAC) will be calculated. This will be expressed as mean difference ± standard deviation in L/min. The ability of EIT to track changes in cardiac output over time will be evaluated by comparing directional changes in CO_EIT with corresponding changes in CO_PAC. This will be reported as the percentage of concordant directional changes between the two methods.
Agreement between EIT-derived and ventilator-measured respiratory parameters | Up to 48 hours
  This outcome assesses the ability of EIT to measure key respiratory parameters compared to the mechanical ventilator measurements. The difference between EIT-derived tidal volume and ventilator-measured tidal volume as well as the difference between EIT-derived respiratory rate and ventilator-measured respiratory rate will be calculated and expressed as mean difference ± standard deviation. Other ventilation-related parameters: Additional parameters such as end-expiratory lung volume changes or regional ventilation distribution may also be assessed, depending on the capabilities of the EIT system and the available ventilator data.

CONTACTS AND LOCATIONS:
Overall Officials: Kaspar F Bachmann, MD, Principal Investigator — Department of Intensive Care Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland; Carmen A Pfortmueller, MD, Study Director — Department of Intensive Care Medicine, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland
Locations (1):
- Inselspital Bern, Universitätsklinik für Intensivmedizin, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No